CLINICAL TRIAL: NCT02167074
Title: A Multicenter Randomized Trial, Comparing a 25G EUS Fine Needle Aspiration (FNA) Device With a 20G EUS ProCore Fine Needle Biopsy (FNB) Device
Brief Title: Comparing a 25G EUS Fine Needle Aspiration (FNA) Device With a 20G EUS
Acronym: ASPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Collaborators: Cook Ireland, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ASPRO-2014-01
Record Dates: First submitted 2014-06-12; First posted 2014-06-18 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Masses; Lymph Nodes
Keywords: Diagnostic accuracy; Endoscopic Ultrasound-Guided Fine Needle Aspiration; EUS-FNA; Endoscopic Ultrasound-Guided Fine Needle Biopsy; EUS-FNB; Pancreatic mass; Lymph node

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 25G FNA needle (Active Comparator): Patients referred for EUS-guided tissue acquisition of a pancreatic mass, lymph node, or other submucosal or undefined mass (non-pancreatic).
  Interventions: Device: 25G FNA needle
- 20G ProCore FNB needle (Active Comparator): Patients referred for EUS-guided tissue acquisition of a pancreatic mass, lymph node, or other submucosal or undefined mass (non-pancreatic).
  Interventions: Device: 20G ProCore FNB needle

INTERVENTIONS:
Device: 25G FNA needle
  Other Names: 25G Echotip Ultra Fine Needle Aspiration (FNA) device
  Arms: 25G FNA needle
Device: 20G ProCore FNB needle
  Other Names: 20G Echotip ProCore Fine Needle Biopsy (FNB) device
  Arms: 20G ProCore FNB needle

SUMMARY:
The aim of this study is to compare the diagnostic accuracy of two EUS-guided tissue acquisition devices; the 25G Echotip Ultra Fine Needle Aspiration (FNA) device and the 20G Echotip ProCore Fine Needle Biopsy (FNB) device.

DETAILED DESCRIPTION:
Endoscopic ultrasound (EUS)-guided tissue acquisition has emerged as a valuable method to diagnose and stage malignancies. During Endoscopic Ultrasound (EUS), tissue samples can be obtained for pathological evaluation with different devices. Fine needle aspiration (FNA) provides a cytological specimen. Unfortunately, in a cytological specimen, inflammatory changes may be undistinguishable from well-differentiated dysplasia. Moreover, for neoplasms such as lymphomas and stromal tumors, tissue architecture and cell morphology are essential for accurate pathological assessment. Therefore, pathologists generally prefer a histological specimen. Fine needle biopsy (FNB) has the advantage of obtaining a histological specimen, which may lead to better diagnostic performance. However, FNB needles are stiffer and more difficult to handle, which can complicate tissue acquisition. In addition, the superiority of histology over cytology in EUS-guided tissue sampling has not been proven yet. For instance, tissue, obtained by FNA and processed with the new cell-block technique, may equal the diagnostic yield of histological tissue cores.

A recent meta-analysis suggested that 25G is the optimal FNA needle size to obtain an adequate cytological specimen. In this study, we aim to compare the properties and merits of a newly designed, more flexible, 20G EUS ProCore FNB device to a conventional 25G EUS-FNA device.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for EUS-guided tissue acquisition because of a (I) pancreatic mass lesion or (II) lymph node
* Age > 18 years
* Written informed consent
* Lesion can be visualized with EUS and is ≥1 cm in size

Exclusion Criteria:

* Known bleeding disorder that cannot be sufficiently corrected with co-fact or fresh frozen plasma (FFP)
* Use of anticoagulants that cannot be discontinued in order to guarantee an INR below 1.5
* Purely cystic lesions
* Previous inclusion in the current study
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco J Bruno, MD, PhD, Study Chair — Erasmus Medical Center; Djuna L Cahen, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (13):
- United States (3):
  - University of California, Irvine, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Stony Brook University Hospital, New York, New York
- The Royal Adelaide Hospital, Adelaide, Australia
- University Hospital Leuven, Leuven, Belgium
- Institut Paoli-Calmettes, Marseille, France
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (2):
  - Vita Salute San Raffaele University, Milan
  - Catholic University Rome, Rome
- Kinki University, Ōsaka-sayama, Japan
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands
- University Hospital of Santiago de Compostella, Santiago de Compostela, Spain
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] van Riet PA, Giorgio Arcidiacono P, Petrone M, Quoc Nguyen N, Kitano M, Chang K, Larghi A, Iglesias-Garcia J, Giovannini M, van der Merwe S, Santo E, Baldaque-Silva F, Bucobo JC, Bruno MJ, Aslanian HR, Cahen DL, Farrell J. Combined versus single use 20 G fine-needle biopsy and 25 G fine-needle aspiration for endoscopic ultrasound-guided tissue sampling of solid gastrointestinal lesions. Endoscopy. 2020 Jan;52(1):37-44. doi: 10.1055/a-0966-8755. Epub 2019 Jul 22. PMID 31330556
- [Derived] van Riet PA, Larghi A, Attili F, Rindi G, Nguyen NQ, Ruszkiewicz A, Kitano M, Chikugo T, Aslanian H, Farrell J, Robert M, Adeniran A, Van Der Merwe S, Roskams T, Chang K, Lin F, Lee JG, Arcidiacono PG, Petrone M, Doglioni C, Iglesias-Garcia J, Abdulkader I, Giovannini M, Bories E, Poizat F, Santo E, Scapa E, Marmor S, Bucobo JC, Buscaglia JM, Heimann A, Wu M, Baldaque-Silva F, Moro CF, Erler NS, Biermann K, Poley JW, Cahen DL, Bruno MJ. A multicenter randomized trial comparing a 25-gauge EUS fine-needle aspiration device with a 20-gauge EUS fine-needle biopsy device. Gastrointest Endosc. 2019 Feb;89(2):329-339. doi: 10.1016/j.gie.2018.10.026. Epub 2018 Oct 24. PMID 30367877

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 patients were included but met exclusion criteria 4 patients were lost to follow-up
Groups:
- 25G FNA Needle: Patients referred for EUS-guided tissue acquisition of a pancreatic mass, lymph node, or other submucosal or undefined mass (non-pancreatic).
  25G FNA needle
- 20G ProCore FNB Needle: Patients referred for EUS-guided tissue acquisition of a pancreatic mass, lymph node, or other submucosal or undefined mass (non-pancreatic).
  20G ProCore FNB needle
Period: Overall Study
Arm/Group | 25G FNA Needle | 20G ProCore FNB Needle
Started | 306 | 302
Completed | 306 | 302
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 25G FNA Needle | 20G ProCore FNB Needle | Total
Number analyzed (Participants) | 306 | 302 | 608
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (0.7) | 66 (0.7) | 66 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 140 | 264
  Male | 182 | 162 | 344
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy
Description: Diagnostic accuracy is the number of correctly diagnosed cases as compared to gold standard diagnosis
  Gold standard diagnosis is defined as;
  1. in operated patients; based on the surgical resection specimen
  2. in non-operated patients; based on the conclusions of the diagnostic work-up (combined outcomes of tissue sampling and imaging studies), and confirmed by a compatible clinical disease course of at least 9 months
Time Frame: 27 months
Measure: Count of Participants; unit: Participants
Arm/Group | 25G FNA Needle | 20G ProCore FNB Needle
Number analyzed (Participants) | 306 | 302
Participants | 237 | 263

2. Secondary Outcome: Number of Participants in Whom Target Lesion Was Sampled
Description: records if a target lesion was reached during the procedure using the randomised needle or not
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | 25G FNA Needle | 20G ProCore FNB Needle
Number analyzed (Participants) | 306 | 302
Participants | 306 | 298

3. Secondary Outcome: Presence of Vital Target Cells Per Case, Per Needle Type
Description: Presence of sufficient vital target cells, as in, target organ cells to provide a diagnosis (yes or no)
Time Frame: after 27 months
Measure: Count of Participants; unit: Participants
Arm/Group | 25G FNA Needle | 20G ProCore FNB Needle
Number analyzed (Participants) | 306 | 302
Participants | 248 | 263
Statistical Analysis 1: Comparison: 25G FNA Needle vs 20G ProCore FNB Needle; Test type: Other — The chi-square test (with Yates' correction when appropriate) or the Fisher exact test was used to compare the two needle types; p < 0.05, Chi-squared

4. Secondary Outcome: Number of Patients With Adverse Events Per Needle Type
Description: adverse events per needle type, up to 27 months after procedure
Time Frame: 27 months after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | 25G FNA Needle | 20G ProCore FNB Needle
Number analyzed (Participants) | 306 | 302
Participants | 3 | 2

5. Secondary Outcome: Diagnostic Yield of the First Needle Pass
Description: Yield is expressed as sample sufficiency for diagnostic analysis by pathologists, this was either sufficient or not
Time Frame: after 27 months
Population: Yield is expressed as sample sufficiency for diagnostic analysis by pathologists, this was either sufficient or not
Measure: Count of Participants; unit: Participants
Arm/Group | 25G FNA Needle | 20G ProCore FNB Needle
Number analyzed (Participants) | 306 | 302
Participants | 206 | 209

6. Secondary Outcome: On-site Pathological Evaluation Performed
Description: Presence of pathologist on site during procedure
Time Frame: 27 months
Measure: Number; unit: participants
Arm/Group | 25G FNA Needle | 20G ProCore FNB Needle
Number analyzed (Participants) | 306 | 302
participants | 74 | 26

ADVERSE EVENTS:
Time Frame: 27 months
Description: it does not differ, 5 adverse events
Arm/Group | 25G FNA Needle | 20G ProCore FNB Needle
All-Cause Mortality (participants affected / at risk) | 0/306 | 0/302
Serious Adverse Events (participants affected / at risk) | 0/306 | 0/302
Other Adverse Events (participants affected / at risk) | 3/306 | 2/302
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 25G FNA Needle (N=306) | 20G ProCore FNB Needle (N=302)
pancreatitis (Gastrointestinal disorders) | 2 | 1
pain (General disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-10-13): https://cdn.clinicaltrials.gov/large-docs/74/NCT02167074/Prot_000.pdf
  • Statistical Analysis Plan (2014-10-13): https://cdn.clinicaltrials.gov/large-docs/74/NCT02167074/SAP_001.pdf